CLINICAL TRIAL: NCT02231138
Title: Efficacy and Safety of Abelmoschus Manihot for Chronic Kidney Disease：a Multicentre Open Study
Brief Title: Efficacy and Safety of Abelmoschus Manihot for Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Jiangsu Suzhong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiangmei Chen, professsor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2014-040-01
Record Dates: First submitted 2014-08-30; First posted 2014-09-04 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Kidney Disease
Keywords: Abelmoschus manihot; Chronic Kidney Disease; proteinuria; efficacy; safety
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abelmoschus manihot (AM) (Experimental): * age above 12 years old (including 12)：huangkui capsule are given orally at 2.5 g three times per day
  * age between 6-12 years old(including 6):huangkui capsule are given orally at 1.5 g three times per day
  * age under 6 years old：huangkui capsule are given orally at 1.0 g three times per day
  Interventions: Drug: Abelmoschus manihot (AM)

INTERVENTIONS:
Drug: Abelmoschus manihot (AM) — Abelmoschus manihot (AM): Huanghui capsule (Jiangsu Suzhong Pharmaceutical Group Co., Ltd.), 0.5 g × 30 capsules/box. A huangkui capsule is a single plant drug extract of Flos Abelmoschus manihot.
  Other Names: Huanghui capsule

SUMMARY:
Huangkui Capsule is a single medicament of traditional Chinese medicine consists of Abelmoschus manihot and has been widely used to treat kidney disease. The purpose of this study is to evaluate the safety and efficacy of Abelmoschus manihot for treating chronic kidney disease in large scale samples with long time take.

DETAILED DESCRIPTION:
The test has not been completed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed as non-ESRD chronic kidney disease (stage I-IV)
* Blood pressure of ≤140/90mmHg
* Obtaining the signed informed consent from patients

Exclusion Criteria:

* Be allergic to Huangkui Capsule
* Combined with severe primary diseases of heart, brain, liver and hematopoietic system and so on, or other serious diseases which can affect the patient's life
* Lactation, pregnancy or plans pregnancy during the study period
* Participating in another clinical study in the same period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in 24-h proteinuria from baseline after treatment | Baseline(week 0), week 12, week 24

SECONDARY OUTCOMES:
change in the serum creatinine level from baseline after treatment | Baseline(week 0), week 12, week 24
change in the estimated glomerular filtration rate (eGFR) from baseline after treatment | Baseline(week 0), week 12, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, MD.& Ph.D, Principal Investigator — Chinese PLA General Hospital
Locations (78):
- China (78):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Military General Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Dong Zhi Men Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - PLA Air Force General Hospital, Beijing, Beijing Municipality
  - PLA Navy General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of General Hospital of PLA, Beijing, Beijing Municipality
  - The Second Artillery General Hospital Of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Xin Qiao Hospital Of Third Military Medical University, Chongqing, Chongqing Municipality
  - Chinese People's Liberation Army No.180 Hospital, Quanzhou, Fujian
  - Chinese People's Liberation Army No.174 Hospital, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - Guizhou Province Hospital of Traditional Chinese Medicine, Guiyang, Guizhou
  - The Affiliated Baiyun Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zun Yi Medical College, Zunyi, Guizhou
  - Hainan Medical College Affiliated Hospital, Haikou, Hainan
  - Hainan Provincial Nong Ken Hospital, Haikou, Hainan
  - Affiliated Hospital of Cheng De Medical College, Chengde, Hebei
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Heilongjiang Provincial Academy of Traditional Chinese Medicine, Haerbin, Heilongjiang
  - The First Affiliated Hospital Of Heilongjiang University of Chinese Medicine, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science And Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huang Gang Central Hospital, Huanggang, Hubei
  - Hubei Provincial Hospital Of TCM, Wuhan, Hubei
  - Union Hospital Tong Ji Medical College Hua Zhong University Of Science And Technology, Wuhan, Hubei
  - Wuhan Integrated TCM & Western Medicine Hospital, Wuhan, Hubei
  - The Second Xiang Ya Hospital of Central South University, Changsha, Hunan
  - Xiang Ya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - Taizhou Traditional Chinese Medicine Hospital, Taizhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Chinese People's Liberation Army No.94 Hospital, Nanchang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The Second Hospital Of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital Of Dalian Medical University, Dalian, Liaoning
  - First Affiliated Hospital of Liaoning Medical University, Jinzhou, Liaoning
  - The General Hospital Of Shenyang Military Region, Shenyang, Liaoning
  - Ningxia Hui Autonomous Region's Hospital, Yinchuan, Ningxia
  - Jinan General Hospital of PLA, Jinan, Shandong
  - Qi Lu Hospital of Shandong University, Jinan, Shandong
  - Jining No.1 People's Hospital, Jining, Shandong
  - Chinese People's Liberation Army No.88 Hospital, Taian, Shandong
  - Yantai Yu Huang Ding Hospital, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Chang Hai Hospital of the Second Military Medical University, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Ren Ji Hospital of Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital Affiliated Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shu Guang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanxi Hospital of Integrated Traditional And Western Medicine, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - The third People's Hospital of Chengdu, Chengdu, Sichuan
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The Second Hospital Of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Hospital of ITCWM, Nankai Hospital, Tianjin, Tianjin Municipality
  - The First Hospital of Shi He Zi Medical University, Shihezi, Xinjiang
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
The test has not been completed.

REFERENCES:
- [Background] Zhang L, Li P, Xing CY, Zhao JY, He YN, Wang JQ, Wu XF, Liu ZS, Zhang AP, Lin HL, Ding XQ, Yin AP, Yuan FH, Fu P, Hao L, Miao LN, Xie RJ, Wang R, Zhou CH, Guan GJ, Hu Z, Lin S, Chang M, Zhang M, He LQ, Mei CL, Wang L, Chen X. Efficacy and safety of Abelmoschus manihot for primary glomerular disease: a prospective, multicenter randomized controlled clinical trial. Am J Kidney Dis. 2014 Jul;64(1):57-65. doi: 10.1053/j.ajkd.2014.01.431. Epub 2014 Mar 14. PMID 24631042